CLINICAL TRIAL: NCT02484742
Title: Pain Sensitization and Habituation in a Model of Experimentally-induced Insomnia Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Monika Haack, Assistant Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2014P000354
Record Dates: First submitted 2015-06-16; First posted 2015-06-30 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Sleep Control Condition; Insomnia Symptoms Induction Condition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep control condition (No Intervention): 8 hours of sleep throughout the 18-day stay in the Clinical Research Center
- Insomnia symptom induction condition (Experimental): 4 4-day cycles, each consisting of 3 nights with sleep disruption followed by one night of recovery sleep.
  Interventions: Behavioral: Insomnia symptom induction

INTERVENTIONS:
Behavioral: Insomnia symptom induction — Several nights during the 18-day stay will be disrupted, such that we delay sleep onset, advance sleep off set, and the sleep period will be disrupted by frequent nighttime awakenings.
  Arms: Insomnia symptom induction condition

SUMMARY:
The main purpose of this study is to learn about the effects of repeated exposure to sleep disruption (3 cycles of sleep disruption, each consisting of three days in a row where sleep is shortened and disrupted, followed by a single night of recovery sleep) on inflammation, mood, and pain processing (experiences/perceptions of pain). Purpose of this research project is to understand the mechanisms of how sleep disruption may change mood and the experience of pain. Understanding those mechanisms is important to develop interventions that may help to reduce the effects of sleep disruption on mood and pain.

DETAILED DESCRIPTION:
1. Screening Procedures: For this research study, the screening procedures include the following activities. Participants will first complete questionnaires and have an interview where they will be asked questions concerning general health status and sleep-wake habits. Also during this visit, a study nurse will collect a small blood sample that will be used to test for a number of markers of general health status.

   If it appears that the participant may be eligible for participation, s/he will be introduced to an electronic diary that will be emailed every morning and evening to monitor sleep-wake patterns, mood, pain, and other health-related information.

   Following the medical screening (visit 2), the physician will determine if the participant is eligible to proceed to the overnight sleep study. This consists of sleeping overnight in the laboratory during the usual sleep time.

   Seven days before participation in the in-hospital portion of the study, a member of the study team will ask the participant to follow the study sleep-wake schedule. Sleep will be monitored with an electronic sleep diary and the participant will wear an actigraphy watch, which will help to evaluate sleep and measure the light level exposure before starting the study.
2. Randomization Procedures: Each participant will complete both parts of the study protocol, i.e., the experimental condition (where participants will undergo repeated cycles of sleep disruption, 18 days total in the Clinical Research Center) and the control condition (where participants will have a sleep opportunity of 8 hours every night; 18 days total in the Clinical Research Center).
3. Research Procedures: If a participant qualifies to take part in this research study, s/he will be required to stay in the hospital for two 18 day long research protocols. These protocols will take place at least 2-3 months apart. The experimental protocol includes 3 nights of 8 hour-sleep per night followed by three 4-day cycles, each consisting of 3 nights of shortened and disrupted sleep, followed by a single night of 8 hour recovery sleep. After the last cycle, the participant will have two more nights with 8 hours of sleep per night. In the control protocol, these 18 days will be 8-hour sleep nights.

   During the stay in the hospital, research staff will accompany the participant during all waking times. The staff will help the participant to stay on the schedule, maintain wakefulness, and make sure that equipment is recording properly.

   Both study protocols will begin with two adaptation nights. On the first day of the protocol, the participant will be told the sleep condition to be assigned first: the sleep disruption condition or the sleep control condition.

   During the sleep disruption nights, sleep onset will be delayed by one hour (midnight 12am), and sleep offset (final wake up) will be advanced by one hour (6am). The sleep period (12-6am) will be disrupted hourly by 20 minute long awakenings. During the nighttime periods, the nurse will measure blood pressure and collect a small sample of your saliva. The participant will also be asked to complete tests that assess well-being and cognitive functioning (such as attention, learning).

   After the last day of the third cycle, the participant will have four nights with 8 hours of sleep per night. The participant will be able to leave the research center in the morning after the 18th night.

   During each of the two 18-day stays in the hospital, participants will wear an actigraphy watch on all study days, which will help to evaluate sleep and measure the light level exposure. The participant will also have two blood draws obtained by a simple needle stick on intermittent days. Additionally, during these 24-hour periods, the study team will be collecting sleep recording data (using a polysomnography device over a 24-hour period). Finally, the study team will collect urine samples over the course of this protocol.

   Blood pressure will be measured at frequent intervals through the study. Computerized performance tests will be conducted at frequent intervals through the study. One of the tests involves measurement of reaction time by having participants press a button on a little box. In another performance test the study team will ask the participant to press the right or left mouse button depending on whether the word on the computer screen is printed in the same color or in a different color; this should be done as quickly and as accurately as possible. In addition, we will ask participants to rate well-being at frequent intervals throughout the stay in the Clinical Research Center.

   On several days during the stay in the Clinical Research Center, the investigators will test the perception of pain. During pain testing, the participant will remain in a comfortable chair throughout the testing session. The testing will consist of measures of pain threshold (first feeling of the sensation of pain to a heat or mechanical stimulus), pain tolerance (when the pain sensation feels intolerable), and pain modulation (how the central nervous system can change the perception of pain).
4. Monitoring/Follow-Up Procedures. For this research study, the monitoring/follow-up procedures include meeting with one of the lead members of the study team on the last day of each of the 18-day protocols. During this time, a study team member will discuss the participant's study experience and will give the opportunity to ask any questions concerning the study.

ELIGIBILITY:
Inclusion Criteria:

* Women and men between the ages 18-45 years.
* Body mass index (BMI) between 18.5 and 30 kg/m2.
* For female participants: regular menstrual cycles, no significant discomfort during pre-menses/menses.
* Good quantity/quality sleep
* Blood chemistry in the normal range.

Exclusion Criteria:

* - Active infection/disease.
* History of neurological, chronic pain, immune, cardiovascular, liver/kidney, or metabolic disorder.
* History of psychiatric disorders, including major depressive disorders, bipolar disorders, panic disorders, post-traumatic stress disorders (PTSD), thought disorders, and substance abuse/dependence disorders.
* Sleep disorders
* Pregnant/nursing.
* Regular medication use other than oral contraceptives.
* Donation of blood or platelets 3 month prior to or in-between study arms.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-07; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers | Followed for the duration of the two in-hospital stays, i.e. 2 x 18 days.
  Pro-inflammatory markers including cytokines (IL-6), prostaglandins (PGE2), measured in blood, urine, and saliva
Pain modulation | Followed for the duration of the two in-hospital stays, i.e. 2 x 18 days.
  Sensitivity to heat and pressure pain, capacity to inhibit a painful stimulus when another painful stimuli is applied at the same time

CONTACTS AND LOCATIONS:
Overall Officials: Monika Haack, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Engert LC, Mullington JM, Haack M. Prolonged experimental sleep disturbance affects the inflammatory resolution pathways in healthy humans. Brain Behav Immun. 2023 Oct;113:12-20. doi: 10.1016/j.bbi.2023.06.018. Epub 2023 Jun 25. PMID 37369338
- [Derived] Haack M, Engert LC, Besedovsky L, Goldstein MR, Devine JK, Dang R, Olia K, Molina V, Bertisch SM, Sethna N, Simpson N. Alterations of pain pathways by experimental sleep disturbances in humans: central pain-inhibitory, cyclooxygenase, and endocannabinoid pathways. Sleep. 2023 Jun 13;46(6):zsad061. doi: 10.1093/sleep/zsad061. PMID 36881901

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT02484742/Prot_SAP_000.pdf